CLINICAL TRIAL: NCT01622829
Title: Pilot Study on Physical Activity
Brief Title: Activity on Prescription to Promote Physical Activity in Hospitalized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Kai Schommer, MD, MD, Heidelberg University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: S-602/2011
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Prescriptions; Exercise

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- group1 (Experimental): Usual Physiotherapy, additional: "Prescription for Activity" with a structured fitness program and individual instructions to become more active in the daily living situation
  Interventions: Procedure: "Prescription for Activity" and individual instructions
- group 2 (Experimental): usual Physiotherapy , additional: "Prescription for Activity" without instructions
  Interventions: Other: "Prescription for Activity", without instructions
- group 3 (No Intervention): control, usual physiotherapy
  Interventions: Other: usual physiotherapy

INTERVENTIONS:
Procedure: "Prescription for Activity" and individual instructions — Structured education. "Prescription for Activity". This contains an exercise programme which consists of a 30 minutes muscle strengthening exercises to be performed at home at least three times per week and an endurance sports, chosen by the patient, to be performed at least 2 times per week. Additional the physiotherapists advise them in being more active during their individual daily life ( e.g. using a bike for short distances, regular walking, abandon the lift/escalator).
  Arms: group1
Other: "Prescription for Activity", without instructions — Prescription with exercise programme. "Prescription for activity". This contains an exercise program consisting of 30 minutes of muscle strengthening exercises to be performed at home at least three times per week, the patient also needs to perform in an endurance sport at least two times per week.
  Arms: group 2
Other: usual physiotherapy — physiotherapy, treatment as usual
  Arms: group 3

SUMMARY:
This study tries to improve patient's activity by a "Prescription for Activity" led by physiotherapists in secondary health care setting.

Three groups are compared in regard to their increase of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-75 years
* self-dependent
* walk around at home alone
* German-speaking
* Ability to read and write
* Life expectancy > 6 months
* Stable disease process expected for the next 6 months
* Time spend in hospital: > 3 days, < 4 weeks

Exclusion Criteria:

* Patients suffering from dementia
* Planned participation in rehabilitation
* severe functional limitations that precluded any increase in physical activity
* not living independently

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in levels of physical activity at three months | Baseline, 3 months
  overall activity score measured in MET*h/week assessed by a modified "Recent Physical Activity Questionnaire" (RPAQ) - Change from Baseline in levels of physical activity at 3 months difference

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Sports Medicine, University of Heidelberg, Heidelberg, Germany